CLINICAL TRIAL: NCT04728191
Title: The Effect of Physiotherapy on Dysfunctional Breathing in Children and Adolescents With and Without Asthma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Signe Vahlkvist, Principal Investigator, Kolding Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20200101-b
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Dysfunctional Breathing; Asthma in Children; Asthma
Keywords: Dysfunctional breathing; Asthma in children; Asthma in adolescents; Physiotherapy
MeSH Terms: conditions — Asthma | interventions — Physical Therapy Modalities; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- + asthma + intervention (Experimental): 35 participants with asthma aged 10-17 years, randomized to physiotherapy. The intervention consists of 4 instruction lessons spread over 6 weeks. The participants are instructed in a daily ten-minute-program of breathing exercizes.
  Interventions: Other: Physiotherapy
- + asthma - intervention (Active Comparator): 35 participants with asthma aged 10-17 years, randomized to standard care. Participants are getting advice about dysfunctional breathing by a physician or nurse in the outpatient clinic.
  Interventions: Other: standard care
- - asthma + intervention (Experimental): 35 participants without asthma aged 10-17 years, randomized to physiotherapy. The intervention consists of 4 instruction lessons spread over 6 weeks. The participants are instructed in a daily ten-minute-program of breathing exercizes.
  Interventions: Other: Physiotherapy
- - asthma - intervention (Active Comparator): 35 participants without asthma, which are randomized to standard care. Participants are getting advise about dysfunctional breathing by a physician or nurse in the outpatient clinic.
  Interventions: Other: standard care

INTERVENTIONS:
Other: Physiotherapy — physiotherapeutical instructions and training as described.
  Arms: + asthma + intervention; - asthma + intervention
Other: standard care — Standard care as described.
  Arms: + asthma - intervention; - asthma - intervention

SUMMARY:
The purpose of the study is to investigate the effect of physiotherapeutical instructions on dysfunctional breathing in children and adolescents with or without asthma.

Children and adolescents with dysfunctional breathing, are invited to participate in the intervention study. Participants are stratified by asthma diagnose status and randomized to physiotherapy or standard care. Participants are followed a year after the intervention, to compare the development in asthma control ( if asthma) and quality of life.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effect of physiotherapeutical instructions on dysfunctional breathing in children and adolescents with or without asthma.

All children and adolescents aged 10-17 years, followed in our outpatient clinic with the diagnose of asthma are invited to fulfill the Nijmegen Questionnaire (NQ) and the Asthma Control Questionnaire (ACQ5)

Children and adolescents where asthma was investigated and ruled out are invited to fulfill the NQ.

Data from the electronic patient journal are used as descriptives.

Participants with dysfunctional breathing (NQ >= 23) are invited to participate in the intervention study. Participants are stratified by asthma diagnose status and randomized to physiotherapy or standard care. Participants are followed a year after the intervention, to compare the development in asthma control measured by ACQ5 (if asthma) and quality of life measured by PedsQL.

The effect of physiotherapy is analyzed separately for participants with and without asthma. In addition, primary outcomes are analyzed in a regression model with asthma status, age and sex as explanatory variables.

ELIGIBILITY:
Inclusion Criteria:

Asthma group:

* Asthma diagnosed by lung function tests and/or typical symptoms.
* Treatment with inhaled corticosteroids in minimum 3 months.
* ACQ5 >= 1.5.
* NQ >= 23.

NonAsthma group

* Asthma denied after lung function tests ( exercise challenge or mannitol challenge)
* NQ >= 23.

Exclusion Criteria:

* Other significant cardiopulmonary or muscoluskeletal conditions.
* Complex functional conditions involving other organ systems.
* patients who already had the physotherapeutical intervention before study start.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Asthma Control Questionnaire ( ACQ5) at 6 months. | ACQ is taken at baseline and 6 months after intervention as primary outcome.
  ACQ5 contains 5 questions regarding asthma symptoms. Each question is scored between 0-6 points, where 0 represents very good asthma control and 6 represents poor asthma control. Total ACQ score is calculates as an average of points. ACQ5 is taken by participants with asthma, at visits in the outpatient clinic.
Change from baseline in Pediatric Quality of Life Inventory ( PedsQl) at 6 months | PedsQL is taken at baseline and 6 months after intervention as primary outcome.
  PedsQl consists of 23 questions in 4 segments ( physical functioning, emotions, social interaction, and school activities). Each question is scored from 0 (best) to 4 (worst). The PedsQl questionnairre exists in formats for young children ( not used here), children aged 8-12 years and Teenagers aged 13-18 years. Children and adolescents are answering the age relevant questionnairre at visits in the out patient clinic. The PedsQl score is transformed to a 0-100 scale as follows: 0 =100, 1=75, 2=50, 3=25, 4=0. Health related Quality of life is calculated as a mean of scores. Psychosocial Health summary score is calculated as a mean of scores in the emotional, social and school functioning scales. Physical Health summary score is calculated as physical functioning scale score mean.

SECONDARY OUTCOMES:
Change from baseline in Nijmegen Questionnaire ( NQ) | NQ is taken at baseline and 6 weeks, 6 months and 12 months after intervention.
  NQ consists of 16 questions regarding dysfunctional breathing. Each question is scored between 0-4 points, where 0 is best and 4 is worst.
Change from baseline in Brompton breathing Pattern Assesment Tool ( BBPAT) | BBPAT is taken at baseline and 6 weeks, 6 months and 12 months after intervention.
  BBPAT is a breathing scoring equipment where an observer is scoring the quality of breathing from seven parameters including respiratory rate, respiratory movements, in and expiratory sounds etc. Each parameter is scored from 0 ( best) to 2 ( worst). Total score is calculated between 0-14 point
Number of contacts to the hospital during one year from baseline | from baseline to 12 months after intervention.
  Number of total contacts includes planned visits, extra visits and hospitalisations
Change from baseline in Asthma Control Questionnaire ( ACQ5) at 6 weeks and one year. Change from 6 months in ACQ at 12 months. | ACQ5 is taken at 6 weeks and 12 months after intervention as secondary outcomes.
  ACQ5 contains 5 questions regarding asthma symptoms. Each question is scored between 0-6 points, where 0 represents very good asthma control and 6 represents poor asthma control. Total ACQ score is calculates as an average of points. ACQ5 is taken by participants with asthma in the outpatient clinic at baseline and after 6 weeks, 6 months and 12 months.
Change from baseline in Pediatric Quality of Life Inventory ( PedsQl) at at 6 weeks and one year. Change from 6 months in PedsQl at 12 months. | PedsQl is taken at 6 weeks and 12 months after intervention as secondary outcomes.
  PedsQl consists of 23 questions in 4 segments ( physical functioning, emotions, social interaction, and school activities). Each question is scored from 0 (best) to 4 (worst). The PedsQl questionnairre exists in formats for young children ( not used here), children aged 10-13 years and Teenagers aged 13-18 years. Children and adolescents are answering the age relevant questionnairre at visits in the out patient clinic. The PedsQl score is transformed to a 0-100 scale as follows. 0 =100, 1=75, 2=50, 3=25, 4=0. Health related Quality of life is calculated as mean of scores. Psychosocial Health summary score is calculated as mean of scores in the emotional, social and school functioning scales. Physical Health summary score is calculated physical functioning scale score mean.
The reported use of rescue Beta2 agonist in puffs per week | at baseline and 6 weeks, 6 months and 12 months after intervention.
  The reported use of short acting beta 2 agonist in puffs per week the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Vahlkvist, PhD, Principal Investigator — Kolding Sygehus
Locations (1):
- Signe Vahlkvist, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie published results, after deidentification.
Supporting Information: SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to Open@rsyd.dk.
URL: http://open.rsyd.dk